CLINICAL TRIAL: NCT00964067
Title: Effect of High Intensity Aerobic Interval Training in Cardiac Rehabilitation
Brief Title: Aerobic Interval Training in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HJERTEREHAB2009
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: rehabilitation outcome; cardiac patients; exercise intensity
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treadmill group (Active Comparator): Interval exercise performed on treadmills, supervised
  Interventions: Other: Exercise training
- Exercise groups (Active Comparator): Supervised and organised in groups of ten
  Interventions: Other: Exercise training
- home-based exercise (Active Comparator): Interval training at home, free choice of modality
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Interval training at 90% of max heart rate. Warm-up of 10-15 minutes up to 70% of HRmax, then 4 minutes of exercise at 90%. 3 minutes of active pause between the intervals. Total 45 minutes of exercise. Twice a week.

SUMMARY:
The purpose of the study is to compare home-based aerobic interval training with supervised interval training performed in groups or on a treadmill at the hospital.

DETAILED DESCRIPTION:
Cardiac rehabilitation is usually first offered in hospitals, but there are several studies that show that home-based rehabilitation is equally efficient. How this comes out when exercise is organized as aerobic interval training is not known.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* age over 18
* referred to cardiac rehabilitation
* exercise tolerance demonstrated

Exclusion Criteria:

* severe arrhythmia
* heart failure
* drug abuse
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
VO2peak | baseline, after 12 weeks and after 1 year

SECONDARY OUTCOMES:
quality of life | baseline, 12 weeks and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Støylen, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- St.Olavs University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Aamot IL, Karlsen T, Dalen H, Stoylen A. Long-term Exercise Adherence After High-intensity Interval Training in Cardiac Rehabilitation: A Randomized Study. Physiother Res Int. 2016 Mar;21(1):54-64. doi: 10.1002/pri.1619. Epub 2015 Feb 16. PMID 25689059
- [Result] Aamot IL, Forbord SH, Gustad K, Lockra V, Stensen A, Berg AT, Dalen H, Karlsen T, Stoylen A. Home-based versus hospital-based high-intensity interval training in cardiac rehabilitation: a randomized study. Eur J Prev Cardiol. 2014 Sep;21(9):1070-8. doi: 10.1177/2047487313488299. Epub 2013 Apr 23. PMID 23613224